CLINICAL TRIAL: NCT01340521
Title: FSH and LH Response to Low Dose Clomiphene Citrate in Normally Menstruating Fertile Women
Brief Title: Follicle Stimulating Hormone (FSH) and Luteinizing Hormone (LH) Response to Low Dose Clomiphene Citrate in Normally Menstruating Fertile Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Carol L. Gnatuk, M.D., The Pennsylvania State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 214-91
Record Dates: First submitted 2011-04-18; First posted 2011-04-22 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Infertility
Keywords: Pituitary Hormone Response; Clomiphene Citrate; Follicle Stimulating Hormone; Luteinizing Hormone
MeSH Terms: conditions — Infertility | interventions — Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Clomiphene Citrate — 0, 25, 50 or 100 milligrams daily. Will be taken orally days five through nine of the menstrual cycle.

SUMMARY:
The goal of the study is to quantitatively evaluate pituitary hormone response, follicle stimulating hormone (FSH) and luteinizing hormone (LH), to low doses of clomiphene citrate in normally fertile women.

DETAILED DESCRIPTION:
Empirical use low-dose clomiphene citrate has been advocated by some practitioners to enhance fecundity in women with unexplained infertility. No clinical trials have examined the efficacy of such treatment in the patient population, although certain studies have shown that active ovulation induction can be effective in women with unexplained infertility, and that cycle fecundity is improved for normally cycling women with active ovulation management in a program of artificial insemination. Since clomiphene citrate can have paradoxical effects on fertility through its anti-estrogenic mode of action, the benefit or lack of benefit from treatment with clomiphene citrate in this patient group needs to be evaluated. We aim to establish a dose response of FSH and LH to various low doses of clomiphene citrate in normally cycling women of known fertility, that is women with an intact hypothalamic-pituitary-ovarian-axis. The significance of this information is that it may help to elucidate the mechanism by which low-dose clomiphene citrate may improve fecundity in patients with unexplained infertility as it is currently being used empirically.

ELIGIBILITY:
Inclusion Criteria:

* Normal cycling healthy women with known fertility
* Regular menses every 24 - 35 days
* 18 to 35 years of age
* be within 20% of ideal body weight
* normal TSH, prolactin and mid luteal phase progesterone

Exclusion Criteria:

* Women with Infertility issues
* Irregular menstrual cycles

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 1991-03; Primary Completion 1994-03 (Actual); Study Completion 1994-03 (Actual)

PRIMARY OUTCOMES:
LH Concentration | Outcome measures assessed every month until menses occur for 4 monthly menstrual cycles
  LH will be measured from blood samples of approximately 10 mL from each subject on cycle day 3 and then daily on cycle day 5 through ovulation as determined by urinary LH testing kit and every 3rd day until menses occur.

SECONDARY OUTCOMES:
FSH Concentration | Outcome measures assessed every month until menses occur for 4 monthly menstrual cycles
  FSH will be measured from blood samples of approximately 10mL from each subject on cycle day 3, then daily from cycle day 5 through ovulation as determined by urinary testing kit and every third day until menses occur.

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Gnatuk, M.D., Principal Investigator — a State University Hershey Medical Center /Mayo Clinic when study was conducted
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States